CLINICAL TRIAL: NCT05230888
Title: A Prospective Study of Comprehensive Geriatric Assessment (CGA) in Non-Small Cell Lung Cancer Patients (NSCLC) Undergoing Treatment With Immune Checkpoint Inhibitors.
Brief Title: Comprehensive Geriatric Assessment in Elderly Non-Small Cell Lung Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: Research personnel not recruited
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: V1.1 10.09.2021
Record Dates: First submitted 2022-01-12; First posted 2022-02-09 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: The effect of immunotherapy treatment will be assessed using the comprehensive geriatric assessment (CGA) and vulnerable elders survey (VES-13) in 100 non-small cell lung cancer patients, aged ≥70 years old, receiving immune checkpoint inhibitor (ICI) treatment.
  Interventions: Other: Questionnaires about symptoms

INTERVENTIONS:
Other: Questionnaires about symptoms — The CGA and VES-13 questionnaires will be conducted at baseline. Immune-related adverse events (irAEs) will be investigated at 3 and 6 months using a Patient Knows Best symptom tracker form (local Trust created).

SUMMARY:
Lung cancer is responsible for one of the highest incidences of cancer-related mortality globally, and non-small cell lung cancer (NSCLC) accounts for the biggest subtype of lung cancer. In recent years, the use of immunotherapy has revolutionised the management of NSCLC, with better response rates and survival outcomes reported in the literature, compared to traditional cytotoxic chemotherapy. Despite this, doubts remain regarding the true efficacy of immunotherapy in patients > 75 years old, given that this age subgroup is mis-represented in prospective phase III trials, in terms of numbers and baseline functional status, compared to real-world experience.

Furthermore, the use of immune checkpoint inhibitors (ICIs) is associated with a spectrum of immune-related adverse events (irAEs), affecting a range of organ systems. Once again, there are doubts about the safety of the use of these agents in patients > 75 years old, and whether baseline performance status and comorbidities are good predictors of efficacy and safety outcomes in this elderly patient subgroup.

Comprehensive Geriatric Assessment (CGA) and the vulnerable elders survey (VES-13) are assessment tools that provide a good indication of functional status in elderly patients, in a similar capacity to performance status and comorbidities. This study therefore aims to prospectively examine patients > 70 years old with a diagnosis of NSCLC, commencing immunotherapy. It will assess CGA and VES-13 scores at baseline, and correlate this with certain outcomes such as the incidence of severe adverse effects from immunotherapy at 3 and 6 months, any admissions to hospital arising from immunotherapy toxicities (and the subsequent length of inpatient stay), and mortality within 30 days. In doing so, it will help to determine if CGA and VES-13 scores can be used as a reliable indication of possible future efficacy and toxicity outcomes in this elderly patient subgroup.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥70 years old with advanced NSCLC due to start first or second line ICI therapy.
2. Patients able to give informed consent.

Exclusion Criteria:

1. Patients already on treatment with ICIs.
2. Patients with CNS or leptomeningeal spread / disease progression.
3. ECOG performance status III/IV.
4. Patients with severe autoimmune diseases.
5. Patients who are recruited and then stop treatment after receiving ≤3 cycles of ICI therapy, secondary to disease progression.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: NSCLC patients ≥70 years old receiving ICI treatment at the Queen's Centre for Oncology and Haematology, Hull.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of irAEs at 3 months. | At 3 months after entering the study.
Nature of irAEs at 3 months. | At 3 months after entering the study.
Grading of irAEs at 3 months. | At 3 months after entering the study.
Incidence of irAEs at 6 months. | At 6 months after entering the study.
Nature of irAEs at 6 months. | At 6 months after entering the study.
Grading of irAEs at 6 months. | At 6 months after entering the study.

SECONDARY OUTCOMES:
Incidence of re-admission into hospital at 3 months. | At 3 months after entering the study.
Incidence of re-admission into hospital at 6 months. | At 6 months after entering the study.
Duration of inpatient stay (conditional on re-admission into hospital). | Up to 12 months after entering the study.
Death within 30 days (if applicable). | Within 30 days of entering the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital, Cottingham, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No